CLINICAL TRIAL: NCT04454567
Title: A Phase 2a, Multi-Center, Single-Blind, Placebo-Controlled Study Evaluating Treatment Intensification With ABI-H0731 in Subjects With Chronic Hepatitis B Infection on Nucleos(t)Ide Reverse Transcriptase Inhibitors
Brief Title: A Study Evaluating Treatment Intensification With ABI-H0731 in Participants With Chronic Hepatitis B Infection on Nucleos(t)Ide Reverse Transcriptase Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to a change in the Sponsor's overall development strategy from treatment of chronic disease to finite, curative treatments, and is based partially on the advice and feedback from experts and regulators.
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-H0731-205; UTN 1111-1251-7136 (Other: World Health Organization)
Record Dates: First submitted 2020-06-18; First posted 2020-07-01 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABI-H0731 + SOC NrtI (Experimental): Participants with chronic hepatitis B virus (HBV) infection with partial virologic suppression on NrtI alone will receive ABI-H0731 300 mg once daily plus standard of care (SOC) NrtI for 96 weeks, followed by SOC NrtI alone for an additional 24 weeks (120 weeks total).
  Interventions: Drug: ABI-H0731; Drug: NrtI
- Placebo + SOC NrtI (Placebo Comparator): Participants with chronic HBV infection with partial virologic suppression on NrtI alone will receive placebo to ABI-H0731 once daily plus SOC NrtI for 48 weeks, followed by ABI-H0731 300 mg once daily plus SOC NrtI for Weeks 48 to 96, followed by SOC NrtI alone for Weeks 96 to 120.
  Interventions: Drug: ABI-H0731; Drug: Placebo; Drug: NrtI

INTERVENTIONS:
Drug: ABI-H0731 — Participants will receive ABI-H0731 tablets orally once daily
Drug: Placebo — Participants will receive placebo to ABI-H0731 tablets orally once daily
  Arms: Placebo + SOC NrtI
Drug: NrtI — Entecavir (ETV), tenofovir alafenamide (TAF), or tenofovir disoproxil fumarate (TDF) SOC according to the respective package insert
  Other Names: Nucleos(t)ide reverse transcriptase inhibitor

SUMMARY:
This study will explore the safety and antiviral activity of ABI-H0731 when added to a nucleos(t)ide reverse transcriptase inhibitor (NrtI) in participants who are partially virologically suppressed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 36 kg/m^2 and a minimum body weight of 45 kg (inclusive)
* In good general health except for chronic hepatitis B (CHB)
* HBeAg positive or HBeAg negative chronic hepatitis B
* HBV DNA >LLOQ using a commercially available assay with LLOQ=20 IU/mL
* On a stable NrtI regimen (ETV, TDF or TAF) for more than 12 months
* Lack of cirrhosis or advanced liver disease

Exclusion Criteria:

* Current or prior treatment for CHB with lamivudine, telbivudine, adefovir, HBV core inhibitor, or previous treatment with an investigational agent for HBV infection
* Presence of substitutions in the HBV polymerase coding region which may confer reduced susceptibility to NrtIs
* Co-infection with human immunodeficiency virus, hepatitis A virus, hepatitis C virus, hepatitis E virus, or hepatitis D virus
* Females who are lactating or wish to become pregnant during the course of the trial
* History or evidence of advanced liver disease or hepatic decompensation
* Clinically significant cardiac disease including poorly-controlled or unstable hypertension; pulmonary disease; chronic or recurrent renal or urinary tract disease; liver disease other than CHB; endocrine disorder; autoimmune disorder; poorly controlled diabetes mellitus; neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment; ongoing infection or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that, in the opinion of the Investigator or the Sponsor, makes the subject unsuitable for trial participation
* History of hepatocellular carcinoma (HCC)
* Exclusionary laboratory parameters at Screening:

  * Platelet count <100,000/mm^3
  * Albumin <lower limit of normal
  * Total bilirubin >1.2 × upper limit of normal (ULN)
  * Direct bilirubin >1.2 × ULN
  * ALT >10 × ULN
  * Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at Screening is >ULN but <100 ng/mL, the participant is eligible if a hepatic imaging trial prior to initiation of study drug reveals no lesions indicative of possible HCC.
  * International Normalized Ratio >1.5 × ULN
  * Glomerular filtration rate <50 mL/min/1.73 m^2 by Chronic Kidney Disease Epidemiology Collaboration equation
  * Any other laboratory abnormality deemed clinically significant by the Sponsor or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knox, Study Director — Assembly Biosciences
Locations (12):
- United States (9):
  - Asia Pacific Liver Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Research and Education, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Schiff Center for Liver Disease, Miami, Florida
  - Institute of Human Virology, Baltimore, Maryland
  - Infectious Disease Care, Hillsborough, New Jersey
  - Northwell Health, Manhasset, New York
  - Office of X.M., MD, Philadelphia, Pennsylvania
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Auckland Clinical Studies, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study Terminated by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 1 | 0 | 1
  United States | 0 | 1 | 1
Years positive for HBV [Mean (Standard Deviation); unit: years] | 4.6 | 45 | 24.8 (28.567)
Years on HBV treatment at Baseline [Mean (Standard Deviation); unit: years] | 3.6 | 1.5 | 2.55 (1.485)
Baseline HBV DNA (Cobas log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 2.20 | 2.06 | 2.13 (0.099)
Baseline HBV pgRNA (log10 U/mL) [Mean (Standard Deviation); unit: log10 U/mL] | 4.85 | 6.55 | 5.7 (1.202)
Baseline HBeAg (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 2.35 | 2.82 | 2.585 (0.332)
Baseline HBcrAg (log10 kU/mL) [Mean (Standard Deviation); unit: log10 kU/mL] | 0.89 | 0.92 | 0.905 (0.021)
Baseline HBsAg (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 3.81 | 4.61 | 4.21 (0.566)
Baseline ALT (U/L) [Mean (Standard Deviation); unit: U/L] | 16 | 11 | 13.5 (3.536)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Time Frame: Baseline and up to 5 months
Measure: Number; unit: participants
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 1 | 1
participants | 0 | 1

2. Primary Outcome: Number of Participants With Premature Discontinuation of Treatment
Time Frame: Baseline and up to 5 months
Measure: Number; unit: participants
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

3. Primary Outcome: Number of Participants With a Laboratory Abnormality
Time Frame: Baseline and up to 5 months
Measure: Number; unit: participants
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

4. Primary Outcome: Number of Participants With HBV DNA <Lower Limit of Quantification (LLOQ) at Week 48
Time Frame: Week 48
Population: Due to early termination of the study, data for Week 48 were not collected and analyzed.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Change From Baseline in log10 HBV DNA
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With HBV DNA <LLOQ at Each Timepoint
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not available to analyze the secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With HBV DNA <Limit of Detection (LOD)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Change From Baseline in log10 HBV Pregenomic RNA (pgRNA)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With HBV pgRNA <LLOQ
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Change From Baseline in log10 Serum Hepatitis B 'e' Antigen (HBeAg)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Change From Baseline in log10 Serum Hepatitis B Core-related Antigen (HBcrAg)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mean Change From Baseline in log10 Serum Hepatitis B Surface Antigen (HBsAg)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Normalized Alanine Aminotransferase (ALT)
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Plasma Concentrations of ABI-H0731
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Plasma Concentrations of Entecavir
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Incidence of HBV Variants Among Participants With Evidence of Non-response to Treatment
Time Frame: Baseline and up to 5 months
Population: Due to early termination of the study, data were not analyzed for secondary outcomes.
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline and up to 5 months
Arm/Group | ABI-H0731 + SOC NrtI | Placebo + SOC NrtI
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-H0731 + SOC NrtI (N=1) | Placebo + SOC NrtI (N=1)
COVID-19 (Infections and infestations) | 0 | 1 (1) — COVID-19 infection
Flu like symptoms (Injury, poisoning and procedural complications) | 0 | 1 (1) — Flu like symptoms secondary to COVID vaccine

LIMITATIONS AND CAVEATS:
Study ABI-H0731-205 was terminated early by the study Sponsor for strategic reasons to prioritize research and development efforts on finite and curative HBV therapies. At the time of early termination, only 2 participants were enrolled, both of which discontinued their assigned study treatment early due to the study being terminated early by the Sponsor. As a result, the primary outcome of number of participants with HBV DNA <LLOQ at Week 48 could not be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Assembly Biosciences agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Assembly Biosciences supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT04454567/Prot_SAP_000.pdf